CLINICAL TRIAL: NCT03799068
Title: Comparative Study of Bilateral Suprazygomatic Maxillary Nerve Block and Surgical Site Infiltration for Perioperative Analgesia in Children Undergoing Cleft Palate Repair
Brief Title: Suprazygomatic Nerve Block vs Surgical Site Infiltration in Cleft Palate Repair
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Maha Nasser Abdellatif Elshimy, Clinical physician, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Cleft Palate
Record Dates: First submitted 2018-11-27; First posted 2019-01-10 (Actual); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Cleft Palate Children; Block
Keywords: bupivacaine; suprazygomatic nerve block
MeSH Terms: conditions — Bites and Stings

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- suprazygomatic maxillary nerve block (Active Comparator): the group were given a bilateral suprazygomatic maxillary nerve block with 0.125% bupivacaine, 2 ml on each side, the total dose of bupivacaine not exceeding 2 mg/kg.
  Interventions: Other: suprazygomatic maxillary nerve block
- surgical site infiltraion (Active Comparator): the group were given peri-incisional infiltration with 0.125% bupivacaine, 2 ml on each side. In all cases the block was given by the anaesthetist and the infiltration by the surgeon.
  Interventions: Other: surgical site infiltration

INTERVENTIONS:
Other: suprazygomatic maxillary nerve block — bilateral Suprazygomatic maxillary nerve block is performed before surgery in anaesthetized children, after aseptic preparation of the skin. The patient is in supine position with the head in neutral position. The puncture site is at the frontozygomatic angle, at the junction of the upper edge of the zygomatic arch and the frontal process. A 24G needle is attached to a syringe containing the local anaesthetic. It is advanced to reach the greater wing of sphenoid at approximately 20 mm depth, then withdrawn a few millimetres and redirected toward the nasolabial fold in a 20° forward and 10° downward direction. The progression in the pterygopalatine fossa is 35 to 45 mm. Loss of resistance after passing through the temporalis muscle assisted in determining the puncture depth. After a negative blood aspiration test, the calculated dose of the local anaesthetic is injected on each side.
  Arms: suprazygomatic maxillary nerve block
Other: surgical site infiltration — peri-incisional infiltration of bupivacaine around the incision site given by the surgeon on an anesthetized patient before the incision is done.
  Arms: surgical site infiltraion

SUMMARY:
The aim of this study is to evaluate the efficacy and duration of effect of bupivacaine given preoperatively as a bilateral suprazygomatic maxillary nerve block and to compare it with peri-incisional infiltration with the same agent for perioperative analgesia in children undergoing cleft palate repair.

DETAILED DESCRIPTION:
Congenital cleft palate (CP) occurs in children at a rate of about 1.5 per 10 000 births, Early surgery is necessary to reduce phonation and feeding difficulties and reduce complications such as frequent sinusitis and other respiratory tract infections. The surgical procedure can be complicated by airway obstruction and respiratory complications. CP is painful in the first 24-48 h following surgery.

Different treatment modalities have been used for reducing or ameliorating the pain following cleft palate repair. These include opioids, paracetamol, non steroidal anti-inflammatory drugs (NSAIDs), surgical site infiltration and various nerve blocks However, the analgesic drugs may provide inadequate analgesia and have side effects such as respiratory depression and bleeding. The inherent disadvantages of analgesic pharmacotherapy in children promoted interest in nerve blocking techniques for operative analgesia. These became established in paediatric anaesthetic practice with the accumulating evidence of advantages such as postoperative pain relief, reduced use of potent narcotics, rapid return of alertness, early feeding and moving about, and early discharge in day care surgery.

The maxillary nerve, the second division of the trigeminal nerve, leaves the cranial part of the face through the foramen rotundum, and then passes forward and laterally through the pterygopalatine fossa, at the bottom of the pterygomaxillary fossa, and reaches the floor of the orbit by the infra- orbital foramen. This sensory nerve supplies innervation of the lower eyelid, the upper lip, the skin between them, the roof of the mouth, and the palate.

Maxillary nerve block through the infrazygomatic route, used for the treatment of trigeminal neuralgia in adults, permits anesthesia of the entire palatine territory. However, this nerve block has lead to complications such as orbital puncture, intracranial injection, maxillary artery puncture, or posterior pharyngeal wall injury In adults, approach to the suprazygomatic MN block (SMB) seems to minimize the risks of the infrazygomatic route providing effective anaesthesia of the entire sensory territory of the MN and its terminal branches.

Bupivacaine, a long-acting amide local anaesthetic has been used widely in infants, particularly for infiltration of wound-edges and nerve blocking.

Pre-incisional infiltration of local anaesthetics has been used both in adults and children in a variety of surgeries with variable results. submucosal infiltration performed by the surgeon seems to alter surgical conditions. Maxillary nerve block using the suprazygomatic approach has demonstrated beneficial effects in adults for trigeminal neuralgia.

ELIGIBILITY:
Inclusion Criteria:

* ASA grade I-III.
* Aged from1-5 years
* Undergoing cleft palate repair.

Exclusion Criteria:

* Patient's refusal.
* Allergy to local anaesthetics.
* Trigeminal neuralgia.
* Bleeding diathesis.
* Inflammation or infection over injection site.

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-03 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Pain assessment | 24 hours postoperative
  By Children's Hospital of Eastern Ontario Pain Scale (CHEOPS) in Young Children (1-7 years) is a behavioral scale for evaluating postoperative pain in young children.
  Cry No crying +1 Moaning,crying +2 Screaming+3
  Facial expression: Smiling +1 Composed, neutral +2 Grimace +3
  Verbal responses Positive statements +1 Negative statement +2 Suffering from pain +3
  Torso Neutral/resting +1 Shifting, shivering, upright +2 Restrained +3
  Legs Neutral position+1 Squirming/kicking, drawn up, tensed legs +2 Restrained +3 Cheops score of 4 or less indicates no pain. Rescue analgesic consisting of paracetamol 10-15 mg/kg will be given rectally when CHEOPS is > 4.

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No